CLINICAL TRIAL: NCT06167928
Title: Investigating the Potential for Musculoskeletal Tissues and Cells Isolated From Juvenile Patients in the Development of Novel Therapies for Cartilage and Bone Injury and Osteoarthritis
Brief Title: Developing Allogeneic Musculoskeletal Therapies
Status: Recruiting | Type: Observational
Sponsor: Keele University (Other)
Collaborators: Alder Hey Children's NHS Foundation Trust (Other); Birmingham Women's and Children's NHS Foundation Trust (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Royal National Orthopaedic Hospital NHS Trust (Other); Scottish National Blood Transfusion Service (Unknown); NHS Blood and Transplant (Other Government); University of Birmingham (Other); Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government); The Royal Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RG-0245-17-ISTM; 21157 (Other Grant/Funding Number: Versus Arthritis); MR/5015167/1 (Other Grant/Funding Number: MRC); 225835 (Other: Health Research Authority (HRA) UK); 17/NW/0550 (Other: REC - North West - Liverpool East)
Record Dates: First submitted 2023-11-21; First posted 2023-12-13 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
Keywords: Cell therapy; Musculoskeletal; Allogeneic
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The bone and cartilage tissue samples will be anonymised and given a unique laboratory number. Any identifiable data (which links the patient to this laboratory number) will be accessible only by the named investigators as a hard copy in a locked storage facility and electronically on a password protected system which complies with the NHS IT security policy. Cells may be isolated from tissues and culture expanded in the laboratory. Cells and tissues will be appropriately stored either at -80 degrees Celsius or in liquid nitrogen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to analyse the cartilage and bone forming potential of cells isolated from the tissues of patients undergoing surgery for the treatment of polydactyly, hip dislocation and from other bio-banked cartilage tissues. The main question it aims to answer is:

Which of the following tissues from polydactyly digit, iliac apophysis or other bio-banked cartilage produce better cartilage in vitro and in vivo? Participants receiving digit amputation surgery for treatment of polydactyly will be asked to donate the associated waste tissue whilst participants receiving surgery to treat a dislocated hip will be asked to donate an extra small piece of cartilage tissue (approximately 1 gram) from the iliac apophysis. Other tissues for the study will be obtained from those donated to biobanks.

DETAILED DESCRIPTION:
Cartilage and bone injury and osteoarthritis (OA) continues to take its toll on the quality of life of a large proportion of the world's population. Clinicians and scientists at the Robert Jones & Agnes Hunt Orthopaedic Hospital (RJAH) are part of the Versus Arthritis Tissue Engineering Centre. The investigators have a long history of developing innovative cell-based therapies for the treatment of cartilage and bone defects and osteoarthritis, such as, autologous chondrocyte implantation, which is considered a successful treatment for chondral defects.

However, there are potential drawbacks to the use of this procedure to treat larger osteochondral defects that arise in OA. These include the potential shortage of cartilage tissue available in OA patients and the fact that those cells obtained may have phenotypes preventing the reproduction of good quality cartilage. It is therefore favourable to seek a source of cells optimal for osteochondrogenesis for every patient.

To further our studies the investigators wish to collect amputated digits that are removed in the routine treatment of polydactyly. The investigators also intend to study cells isolated from the iliac apophysis, these tissues will be removed during surgeries in the treatment of dislocated hips. In addition, the investigators intend to receive joint tissues from collaborative orthopaedic hospital tissue biobanks and National Health Service Blood and Transplant (NHS-BT). Our intention is to study the potential of cells derived from these tissues in the treatment of other patients with cartilage or bone injuries or osteoarthritis.

In the first instance, the investigators propose to evaluate the use of various sources of cells for musculoskeletal therapies including bone, bone marrow and cartilage, although skin, fat and other tissues might also be attractive sources. Stem cells derived from these tissues are known to be capable of differentiating into cells which might be suitable for musculoskeletal repair strategies, i.e. osteoblasts and chondrocytes, to form bone and cartilaginous tissues. Thus these cells are attractive candidates for allogenic cell therapies for treatment of OA tissue damage. Furthermore the expected high vitality of the juvenile cells may allow for several patients to be treated by one characterised source. This will help to lower the cost of providing a cell therapy.

ELIGIBILITY:
Inclusion Criteria:

For juvenile/infant donors:

* Parents/guardians being able to provide signed and dated informed consent form.
* Scheduled for one of the following surgical treatments:

Digit amputations due to polydactyly. Surgery to treat dislocated hips.

For biobank/NHSBT donors

* Informed consent via consenting institution.

Exclusion Criteria:

* Parents/guardians not understanding the Patient Information Sheet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Juvenile/infant donors:
  Participants between 0-4 years of age scheduled for polydactyly digit amputation or hip dislocation surgeries at the RJAH Orthopaedic, Alder Hey, Norwich and Norfolk, Royal National Orthopaedic and Birmingham Women's and Children's Hospitals (where appropriate i.e. polydactyly only at Alder Hey, and Norwich and Norfolk.
  Biobank/NHSBT donors:
  Participants of any age that have consented to donating their cartilage tissues to a bio-bank.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2037-09-01 (Estimated)

PRIMARY OUTCOMES:
Cell viability as assessed by trypan blue exclusion assay | Up to 48 hours
  The viability of cells post-collagenase digest will be assessed by trypan blue exclusion assay

SECONDARY OUTCOMES:
Measure levels of glycosaminoglycan content by 1,9-dimethylmethylene blue (DMMB) assay | Up to 3 months
  Glycosaminoglycan levels will be measured post-chondrogenic induction by DMMB assay

CONTACTS AND LOCATIONS:
Overall Officials: Karina T Wright, PhD, Principal Investigator — ISTM, Keele University
Locations (1):
- Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust, Oswestry, Shropshrie, United Kingdom

IPD SHARING:
Plan to Share IPD: No